CLINICAL TRIAL: NCT06026956
Title: Validity and Reliability of Fitnessgram and Pediatric Functional Reach Tests Applied With Face-to-Face and Tele-Assessment Methods in Children With Asthma
Brief Title: Tele-Assessment Methods in Children With Asthma
Acronym: TeleAssessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Şeyma Nur Önal, Lecturer, Bartın Unıversity
Other Study IDs: GO23/26
Record Dates: First submitted 2023-08-09; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Asthma Childhood
Keywords: Asthma Childhood; Tele-assessment; Fitness Test; Reach Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tele-Assessment — Tele-Assessment

SUMMARY:
Asthma is a chronic inflammatory disease of the airways. Childhood asthma is quite common. The airway responds unusually to triggers. There are episodes of recurrent wheezing, shortness of breath, chest tightness, and/or coughing that may change in intensity over time. Sudden contraction of airway smooth muscle may be reversible. It is characterized by common but also variable airflow obstruction. With the development of today's technology age, tele-assessment techniques allow professionals to remotely collect real-time data about the development of patients. It has been shown that video conferencing is a feasible and reliable method for evaluating patients with neurological symptoms. In a systematic study examining 41 articles investigating telehealth services and satisfaction; The findings show that patients are generally satisfied with the use of telemedicine. He argues that telemedicine is a low-cost model, increases access to health services, saves time, eliminates the need for travel, facilitates remote patient care and follow-up, and also improves health outcomes and/or quality. Therefore, the aim of our study; To compare the findings obtained with tele-assessment and clinical face-to-face evaluations on a scientific basis, where tele-applications are developing rapidly and their effectiveness has been proven by research, and according to the data to be obtained, an idea about the compatibility between remote evaluation of some parameters of asthmatic children such as physical fitness and flexibility, balance and face-to-face evaluations. is to own. In different situations where patients cannot reach the clinic (remote distance, pandemic, etc.), the evaluations to be made using the remote tele-assessment method can reflect the objective data and the continuity of the patient-health professional relationship can be maintained.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease of the airways. Childhood asthma is quite common. The airway responds unusually to triggers. There are episodes of recurrent wheezing, shortness of breath, chest tightness, and/or coughing that may change in intensity over time. Sudden contraction of airway smooth muscle may be reversible. It is characterized by common but also variable airflow obstruction. Different classifications can be made according to age, symptoms, severity and inflammation in the school and pre-school period. Generally, allergic asthma is common. It is also possible to have atopic dermatitis, allergic rhinitis and food allergy in their personal and family history. In physical examination in children with asthma; They should be carefully examined for signs such as cyanosis, tachycardia, increased air trapping in the lungs, use of auxiliary respiratory muscles, intercostal/suprasternal/subcostal retractions, and difficulty in speaking. The degree of bronchospasm caused by physical activity differs from individual to individual and may vary daily depending on other triggers that the child is exposed to. Mucus accumulation due to the course of the disease, recurrent asthma attacks; It can cause pathological respiratory pattern, posture disorder and circulatory system disorders. In the later stages of the disease, continuous use of accessory respiratory muscles instead of the diaphragm leads to spinal immobility, shortening of the chest muscles, raised and dropped shoulders, forward tilt of the head, and shortening of the muscles around the hips and knees. In the chronic phase, inflammation of the lungs causes the body to deform. These negative physical changes can lead to problems with physical fitness and balance. Physical assessment plays a key role in detecting dysfunctions and activity limitations, establishing the rehabilitation program and determining its effectiveness. With the development of today's technology age, tele-assessment techniques allow professionals to remotely collect real-time data about the development of patients. It has been shown that video conferencing is a feasible and reliable method for evaluating patients with neurological symptoms. In a systematic study examining 41 articles investigating telehealth services and satisfaction; The findings show that patients are generally satisfied with the use of telemedicine. He argues that telemedicine is a low-cost model, increases access to health services, saves time, eliminates the need for travel, facilitates remote patient care and follow-up, and also improves health outcomes and/or quality. Therefore, the aim of our study; To compare the findings obtained with tele-assessment and clinical face-to-face evaluations on a scientific basis, where tele-applications are developing rapidly and their effectiveness has been proven by research, and according to the data to be obtained, an idea about the compatibility between remote evaluation of some parameters of asthmatic children such as physical fitness and flexibility, balance and face-to-face evaluations. is to own. In different situations where patients cannot reach the clinic (remote distance, pandemic, etc.), the evaluations to be made using the remote tele-assessment method can reflect the objective data and the continuity of the patient-health professional relationship can be maintained. The investigators also think that asthmatic children, whose physical evaluations can be made remotely with the data to be obtained, may have advantages such as transportation, weather conditions, school attendance, control of triggers (crowded environments, cigarette smoke, polluted air, etc.). The interviews will be recorded on the computer of the principal investigator and personal data will be recorded in accordance with the Personal Data Protection Law, the law and the rules of honesty, accurate and when necessary, for current, specific, clear and legitimate purposes, in connection with the purpose for which they are processed, limited and measured, for the purpose stipulated in the relevant legislation or for the purpose for which they are processed. Preservation rules will be followed for as long as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Hacettepe University Faculty of Medicine, Department of Pediatrics, Allergy and Asthma Unit patients referred for Cardiopulmonary Rehabilitation,
* Those who have been diagnosed with asthma,
* Clinically stable and not in active asthma attack,
* Between the ages of 6-11,
* Giving consent on a voluntary basis,
* cooperative,
* Ability to use a smart phone or computer,
* Individuals with internet connection will be included in the research.

Exclusion Criteria:

* Individuals with asthma were included in the study.
* Those whose clinical status is not stable and who are in active asthma attack,
* Having serious diseases such as cancers, heart failure and acute respiratory infections,
* Having chronic lung disease other than asthma,
* Severe neuromuscular and musculoskeletal problems,
* Uncooperative to do the tests,
* For safety reasons, patients admitted or hospitalized in the last 3 months due to an asthma attack will not be included in the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthmatic Child
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
FİTNESSGRAM (a)Sit and lie down test with back support: | one day
  The test, which measures physical fitness parameters, can be applied to 5 inpatients. Appropriate cut-off points are specified in the application guide.
  (a)Sit and lie down test with back support: While sitting, the person extends his foot and leans on the bench and bends the other lower extremity. The hands are stretched forward four times in a row and the fourth distance is recorded.
FİTNESSGRAM (b)Trunk Extension-extension test: | one day
  (b)Trunk Extension-extension test: The person lies face down with the hands under the thighs. He lifts his body twice, looking at a coin. In the second, the distance between the chin and the cushion is recorded.
FİTNESSGRAM (c)Trunk Flexion flexion test: | one day
  (c)Trunk Flexion flexion test: The person lies on his back with the knees bent and touches the fixed band on the sides at hand level with the fingertips. Lifts the trunk in a repeat rhythm (every three seconds). It does not move from the lane while rubbing its hands. The number of repetitions performed correctly in accordance with the rhythm is noted.
FİTNESSGRAM (d)Push-up test: | one day
  (d)Push-up test: The person is face down and the hands are shoulder-width apart. The chest moves up and down, with the elbows locked and unlocked (every three seconds) without bending the body. The number of repetitions is noted.
FİTNESSGRAM (e) Progressive aerobic cardiovascular endurance test (PACER): | one day
  (e) Progressive aerobic cardiovascular endurance test (PACER): The set time to reach 20 meters is 9 seconds. If the rhythm cannot be kept up or the boundary line is not reached before the beep twice, the test is stopped, and the number of laps is recorded.

SECONDARY OUTCOMES:
Pediatric Reach Test | one day
  Evaluates the dynamic component of balance. It has validity and reliability for healthy and disabled children. The test is performed by recording the distance, in cm, at which the subjects can reach forward, then to the right and left, respectively, in sitting (with the hip and knee flexed to 90 degrees, in a chair without side and back support) and standing upright positions without lifting their heels off the ground.

IPD SHARING:
Plan to Share IPD: No